CLINICAL TRIAL: NCT06567080
Title: An Open Label, Single Arm Study to Evaluate JWCAR201 Treating B Cell Driven Hematology Malignancy and Autoimmune Diseases
Brief Title: JWCAR201 for the Treatment of Hematology Malignancy and Autoimmune Diseases
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: Shanghai Ming Ju Biotechnology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Liangjing Lu, Professor, RenJi Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JWCAR201001
Record Dates: First submitted 2024-08-15; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: B-cell Tumors; Autoimmune Diseases; Lupus Erythematosus, Systemic; Large B-cell Lymphoma
MeSH Terms: conditions — Autoimmune Diseases; Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JWCAR201 arm (Experimental): Subjects in this arm will receive intervention with JWCAR201
  Interventions: Biological: JWCAR201

INTERVENTIONS:
Biological: JWCAR201 — JWCAR201 is a autologous CAR-T targeting CD19/CD20

SUMMARY:
JWCAR201 is a CD19/CD20 CAR-T product. This trial is intended to evaluate the safety, PK/PD and efficacy of JWCAR201 in patients with B cell driven hematology malignancy and autoimmune diseases

DETAILED DESCRIPTION:
JWCAR201 is a CD19/CD20 CAR-T product. By targeting both CD19 and CD20, it is expected to overcome some limitations with CD19 or CD20 single target products. In this study, patients with B cell driven hematology malignancy and autoimmune diseases will be enrolled to receive JWCAR201. PK/PD properties and preliminary efficacy and safety will be evaluated. Each subject will receive JWCAR201 once and is followed up for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

For subjects with B cell driven malignancy (relapsed/refractory large B cell lymphoma)

1. aged >= 18 years
2. willing to sign ICF
3. with histologically confirmed large B cell lymphoma and immunohistochemically positive CD20
4. The subject must have previously been treated with an anthracycline and rituximab (or another CD20-targeted therapy), and must have relapsed, not achieved remission, or experienced disease progression after receiving at least two lines of therapy, including autologous hematopoietic stem cell transplantation (autoHSCT)
5. The subject must have CT measurable lesions and PET evaluable lesions as determined by the Lugano criteria.
6. The subject must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

For subjects with SLE:

1. Voluntarily sign the informed consent form (ICF).
2. At the time of signing the ICF, be between 18 and 70 years old (inclusive of 18 and 70 years), with no restriction on gender.
3. Have been diagnosed with SLE (Systemic Lupus Erythematosus) for ≥ 6 months before screening, according to the 2019 EULAR/ACR revised criteria
4. Have previously required treatment with corticosteroids combined with immunosuppressants and biologics, with the treatment regimen stable for >2 months and the dose stable for >2 weeks before screening, yet the disease remains active.
5. At the time of screening, positive for antinuclear antibodies (ANA), and/or anti-dsDNA antibodies, and/or anti-Smith antibodies.
6. SLEDAI-2K score ≥ 7 points during the screening period.

   Exclusion Criteria:

   For subjects with B cell driven malignancy (relapsed/refractory large B cell lymphoma)

1. Primary central nervous system (CNS) lymphoma (subjects with secondary CNS lymphoma are allowed to enroll).

2. A history of another malignancy that has not been in complete remission for at least 2 years (the following conditions are exempt from the 2-year restriction: non-melanoma skin cancer, completely resected stage I tumors with a low likelihood of recurrence, treated localized prostate cancer, biopsy-confirmed in situ cervical cancer, or squamous intraepithelial lesions identified on a PAP smear).

3. At the time of screening, the subject has:

1. Hepatitis B surface antigen (HBsAg) positivity (regardless of whether or not there is an increase in hepatitis B virus DNA copies).
2. Hepatitis B core antibody (HBcAb) positivity with an increase in hepatitis B virus DNA copies.
3. Hepatitis C, HIV, or syphilis infection. 4. The subject has had active deep vein thrombosis (DVT) (tumor thrombus or blood clot) or pulmonary embolism (PE) within 3 months prior to signing the informed consent form.

5. The subject has been undergoing anticoagulant therapy for active DVT or PE within 3 months prior to signing the informed consent form (prophylactic treatment is excluded).

6. Uncontrolled systemic fungal, bacterial, viral, or other infections. 7. Acute or chronic graft-versus-host disease (GvHD). 8. History of any of the following cardiovascular diseases within the past 6 months: New York Heart Association (NYHA) Class III or IV heart failure, cardiac angioplasty or stenting, myocardial infarction, unstable angina, or other clinically significant heart diseases.

9. Clinically significant CNS diseases within the past 6 months or at the time of screening, such as epilepsy, seizures, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychiatric disorders.

10. Pregnant or breastfeeding women. Women of childbearing potential must have a negative serum pregnancy test within 48 hours prior to the start of lymphodepleting chemotherapy.

11. The investigator determines that the subject has any factors that could affect compliance with the protocol, including uncontrolled medical, psychological, familial, sociological, or geographical conditions; or the subject is unwilling or unable to comply with the procedures required by the study protocol.

12. The subject has previously received CAR-T cell therapy or other gene-modified T cell therapy.

For subjects with SLE:

1. Severe lupus nephritis requiring hemodialysis within 2 months before screening, or treatment with prednisone ≥ 100 mg/day or equivalent corticosteroids for ≥ 14 days.
2. Lupus crisis within 1 month before screening, deemed unsuitable for participation in this study by the investigator.
3. Clinically significant central nervous system disease or pathological changes not caused by lupus before screening, including but not limited to: cerebrovascular accident, aneurysm, epilepsy, seizures/convulsions, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis. Central nervous system manifestations caused by lupus before screening, including but not limited to lupus headache, seizures, cognitive impairment, intellectual disability, visual impairment, etc.
4. Concurrent other autoimmune diseases requiring systemic treatment.
5. History of major organ transplantation (e.g., heart, lung, kidney, liver) or hematopoietic stem cell/bone marrow transplantation.
6. At the time of screening:

1)Active hepatitis B. 2)Hepatitis C, HIV, or syphilis infection. 7. History of any of the following cardiovascular diseases within 6 months before screening: New York Heart Association (NYHA) Class III or IV heart failure, myocardial infarction, unstable angina, uncontrolled or symptomatic atrial arrhythmias, any ventricular arrhythmias, or other clinically significant heart diseases.

8. Use of any other investigational drug for SLE within 1 month before screening. However, if the investigational treatment was ineffective or the disease relapsed during the study treatment period, and at least 3 half-lives of the drug have passed before screening, the patient may be eligible for enrollment.

9. Previous treatment with CAR-T cells or other gene-modified T cell therapies. 10. History of ≥ Grade 2 bleeding within 30 days before screening, or the need for long-term continuous use of anticoagulant medications (such as warfarin, low molecular weight heparin, or factor Xa inhibitors).

11. Undergoing plasmapheresis, plasma exchange, or hemodialysis within 14 days before screening.

12. Use of any live vaccines for infectious diseases within 1 month before screening.

13. Known life-threatening allergic reaction, hypersensitivity, or intolerance to JWCAR201 cell product or its excipients (including dimethyl sulfoxide (DMSO)).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
the rate of Dose Limiting Toxicity events | 28 days
  Dose-Limiting Toxicity (DLT) refers to a specific type of adverse effect or toxic reaction caused by a drug or treatment that is severe enough to prevent an increase in dose or continuation of treatment.
the rate of AE and SAE | up to 2 years
  any adverse event (AE) or serious adverse event (SAE) occurring after JWCAR201 administration

SECONDARY OUTCOMES:
the change of number of JWCAR201 cells by measuring the cell number and the number of transgene copies over time | from baseline up to 2 years
  to evaluate PK properties of JWCAR201, that is, how the human body processes the infused JWCAR201 cells
the change of numbers of B cell subtypes (e.g., CD19+, CD20+ B cells) in the blood | from baseline up to 2 years
  these are parameters to evaluate PD properties of JWCAR201
overall response rate (ORR) in subjects with hematology malignancy | from baseline up to 2 years
  ORR is the proportion of subjects who achieve positive response to the treatment. It includes complete response and partial response.
complete response rate (CRR) in subjects with hematology malignancy | from baseline up to 2 years
  CRR refers to the proportion of subjects whose cancer signs disappear
duration of response in subjects with hematology malignancy | from baseline up to 2 years
  The duration of a subject staying in response state
progression free survival in subjects with hematology malignancy | from baseline up to 2 years
  the length of time during and after treatment that a subject lives with the disease without the disease worsening or progressing
Overall survival in subjects with hematology malignancy | from baseline up to 2 years
  the length of time from the start of treatment that patients are still alive
the proportion of subjects achieving LLDAS in subjects with SLE | from baseline up to 2 years
  Lupus Low Disease Activity State (LLDAS) is a target for treatment, representing a state where the disease is under control to a degree that is considered acceptable for the patient's long-term health and well-being. It includes below requirements: (1) SLE Disease Activity Index (SLEDAI)-2K ≤4, with no activity in major organ systems (renal, central nervous system (CNS), cardiopulmonary, vasculitis, fever) and no haemolytic anaemia or gastrointestinal activity; (2) no new lupus disease activity compared with the previous assessment; (3) a Safety of Estrogens in Lupus Erythematosus National Assessment (SELENA)-SLEDAI physician global assessment (scale 0-3) ≤1; (4) a current prednisolone (or equivalent) dose ≤7.5 mg daily; and (5) well tolerated standard maintenance doses of immunosuppressive drugs and approved biological agents.
the proportion of subjects achieving DORIS in subjects with SLE | from baseline up to 2 years
  Definitions of Remission in SLE (DORIS) is considered an optimal treatment goal, indicating that the disease is inactive and that the patient has minimal or no symptoms. DORIS includes below requirements: clinical systemic lupus erythematosus disease activity index (SLEDAI)-2K=0, Evaluator's Global Assessment <0.5 (0-3), prednisolone 5 mg/day or less, and stable antimalarials, immunosuppressives, and biologics.
the proportion of subjects achieving SRI-4 in subjects with SLE | from baseline up to 2 years
  Systemic Lupus Erythematosus Responder Index-4 (SRI-4) is a composite index used in clinical trials to assess the effectiveness of treatments for SLE. To be considered a responder according to SRI-4, a patient must meet the following criteria:
  1. Reduction in SLEDAI-2K Score by ≥ 4 Points:
  2. No New BILAG A Scores, and No More Than 1 New BILAG B Score:
  3. No Worsening in Physician's Global Assessment (PGA):
the change of BILAG-2004 score in subjects with SLE | from baseline up to 2 years
  British Isles Lupus Assessment Group (BILAG)-2004 is a score designed to evaluate lupus disease activity across nine organ system. For each organ system, disease activity is assessed and categorized into one of five levels:
  A (Severe Activity): High disease activity requiring significant treatment, such as starting or increasing high-dose immunosuppressive therapy or biologics.
  B (Moderate Activity): Moderate disease activity that might require an increase in treatment, such as adding or increasing corticosteroids or other immunosuppressive drugs.
  C (Mild Activity): Mild disease activity that might not require a change in current treatment.
  D (No Current Activity but Presence of Past Disease): The patient has no current disease activity, but there is evidence of past disease involvement in that organ system.
  E (No Current or Past Activity): The patient has no current or past disease activity in that organ system.
the change of Physician's global assessment (PGA) score in subjects with SLE | from baseline up to 2 years
  PGA is a subjective measure where the physician evaluates and rates the patient's disease activity based on their clinical judgment, considering all aspects of the disease, ranging from 0 to 3. The higher the score, the more severe the disease activity.
the change of SLE-DAS score in subjects with SLE | from baseline up to 2 years
  Systemic Lupus Erythematosus-Disease Activity Score (SLE-DAS) is a validated, continuous measure of disease activity in patients with Systemic Lupus Erythematosus, typically ranging from 0 to over 20. The higher the score, the more active the disease.
the proportion of subjects without other SLE therapies | from baseline up to 2 years
  If JWCAR201 works well, subjects would not need other SLE therapies
The change of fatigue score in subjects with SLE | from baseline up to 2 years
  Fatigue is one of the common symptoms of SLE subjects. A numerical rating scale ranging from 0-10 will be used to assess fatigue, the higher the score, the more severe the fatigue.
The change from baseline in immunoglobulins (IgA, IgE, IgG, IgM) | from baseline up to 2 years
  JWCAR201 can deplete B cells, thus decrease the concentration of immunoglobulins, which are produced by B cells.
the change from baseline in complements (C3, C4) | from baseline up to 2 years
  Complement levels, C3 and C4, increase in active SLE and will decrease following effective treatment
The change from baseline in auto-antibodies (anti-dsDNA antibody, ANA) | from baseline up to 2 years
  anti-dsDNA and ANA antibodies are auto-reactive antibodies produced by pathogenic B cells. JWCAR201 can deplete pathogenic B cells and decrease concentration of the auto-antibodies, indicating the improvement of SLE.

CONTACTS AND LOCATIONS:
Overall Officials: Liangjing Lu, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No